CLINICAL TRIAL: NCT01501409
Title: Effect of Sodium Lauryl Sulfate on Recurrent Aphthous Stomatitis : a Randomised Clinical Trial
Brief Title: Effect of Sodium Lauryl Sulfate on Recurrent Aphthous Stomatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Shim Young Joo, research fellow, Yonsei University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2-2009-0012
Record Dates: First submitted 2011-12-23; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: Sodium lauryl sulfate (SLS); recurrent aphthous stomatitis (RAS); dentifrice; pain
MeSH Terms: conditions — Stomatitis, Aphthous; Pain | interventions — Sodium Dodecyl Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (Experimental)
  Interventions: Other: sodium lauryl sulfate
- Group II (Active Comparator)
  Interventions: Other: sodium lauryl sulfate
- Group III (Active Comparator)
  Interventions: Other: sodium lauryl sulfate

INTERVENTIONS:
Other: sodium lauryl sulfate — The subjects were divided into three groups, each of which comprised 30 randomly assigned subjects: group I used SLS-free(a commercially available SLS-free dentifrice(Wiconi® dentifrice) and SLS-A (a dentifrice containing 1.5%; Wiconi® dentifrice + 1.5% SLS). The subjects used one of the two assigned dentifrices for 8 weeks, and then the other for the following 8 weeks. The order of the dentifrices used was selected at random, and there was a 2-week washout period between the two phases, during which the subject used the same dentifrice as they used before participating in this study. The subjects were asked to brush their teeth using their usual toothbrushing method with the dentifrice and toothbrush supplied.
  Arms: Group I
Other: sodium lauryl sulfate — The subjects were divided into three groups, each of which comprised 30 randomly assigned subjects: group II used SLS-A (a dentifrice containing 1.5%; Wiconi® dentifrice + 1.5% SLS) and SLS-B (a commercially available 1.5% SLS-containing dentifrice). The subjects used one of the two assigned dentifrices for 8 weeks, and then the other for the following 8 weeks. The order of the dentifrices used was selected at random, and there was a 2-week washout period between the two phases, during which the subject used the same dentifrice as they used before participating in this study. The subjects were asked to brush their teeth using their usual toothbrushing method with the dentifrice and toothbrush supplied.
  Arms: Group II
Other: sodium lauryl sulfate — The subjects were divided into three groups, each of which comprised 30 randomly assigned subjects: group III used SLS-free (a commercially available SLS-free dentifrice (Wiconi® dentifrice), and SLS-B (a commercially available 1.5% SLS-containing dentifrice). The subjects used one of the two assigned dentifrices for 8 weeks, and then the other for the following 8 weeks. The order of the dentifrices used was selected at random, and there was a 2-week washout period between the two phases, during which the subject used the same dentifrice as they used before participating in this study. The subjects were asked to brush their teeth using their usual toothbrushing method with the dentifrice and toothbrush supplied.
  Arms: Group III

SUMMARY:
Sodium lauryl sulfate (SLS) is an anionic detergent that has been used as the major or sole surfactant in most dentifrices. But it is known to local irritating factor to oral mucosa and skin and results in many side effects. This study was to compare the effects of SLS-free dentifrice and SLS-containing dentifrice in patients with recurrent aphthous stomatitis (RAS).

ELIGIBILITY:
Inclusion Criteria:

* The volunteers had a history of regularly recurring oral ulcerations of at least 6 months duration, with more than one episode per month

Exclusion Criteria:

* already using an SLS-free dentifrice
* taking medications affecting oral ulcers (e.g., corticosteroids)
* having chronic oral mucosal disease (ex, lichen planus, pemphigus vulgaris, pemphigoid, and etc.)
* having allergies to food or medications
* being pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of episodes | after 18 weeks
  Sum of the number of episodes experienced by the subject over an 8-week period

SECONDARY OUTCOMES:
Mean pain score | after 18 weeks
  Mean pain scores (on the NRS*) experienced during tooth brushing when ulcers were present
  * NRS : numeric rating scale
Number of ulcers | after 18 weeks
  Sum of the number of ulcers over an 8-week period
duration of ulcers | after 18 weeks
  Sum of the number of days which the subject experienced ulcers over an 8-week period

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Seung Kwon, Study Director — Yonsei University dental hospital